CLINICAL TRIAL: NCT04029740
Title: Searching for Exosomal microRNAs and Cellular Biomarkers and Mechanisms Underlying the Differences Between Panic Disorder Patients Who Are Responders and Non-responders to Cognitive Behavior Therapy
Brief Title: Exosomal microRNAs as a Biomarker in Panic Disorder and in Response to CBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebrew University of Jerusalem (Other)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Jonathan D. Huppert, Professor, Hebrew University of Jerusalem
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0577-18-HMO
Record Dates: First submitted 2019-05-22; First posted 2019-07-23 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: All patients will be treated with either internet or face to face CBT according to their preference. Circulating exosomal microRNAs will be measured pretreatment and post-treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy controls (Other): 40 Healthy controls matched on gender and age with no current psychopathology will have exosomal microRNAs measured twice over a 3 month period.
  Interventions: Other: No intervention
- panic disorder receiving CBT (Experimental): 40 adult patients diagnosed with primary panic disorder will have their exosomal microRNAs measured 2x over 3 months.
  Interventions: Behavioral: CBT- both internet and face to face

INTERVENTIONS:
Behavioral: CBT- both internet and face to face — There are a few common psychotherapies for treating PD, with Cognitive Behavioral Therapy (CBT) as the most common. The most known type of CBT for treating PD consists of two major strategies: cognitive restructuring, and interoceptive and structured exposure to bodily sensations that have become associated with panic attacks (D H Barlow, 1997). The ICBT therapy is based on Barlow and Craske's (2007) protocol for treating PD with elaborations (Huppert & Baker-Morissette, 2003). It includes six modules containing psychoeducation, cognitive restructuring, exposures, acceptance, and consolidation of gains and relapse prevention. The online modules include reading passages, worksheets, videos, and homework assignments. After completing each module, participants practice related skills and complete homework assignments. The treatment is up to 16 weeks long; participants are encouraged to complete the treatment within this time period, and reminders are sent to monitor their progress.
  Other Names: Cognitive behavioral therapy for panic disorder
  Arms: panic disorder receiving CBT
Other: No intervention — Healthy controls will not receive any intervention.
  Arms: Healthy controls

SUMMARY:
Cognitive behavior therapy (CBT) has long been known as an effective treatment for anxiety disorders, either when given by a therapist or when self-administered through a computer program. However, the biological effect of CBT remained largely unexplored. Most studies focused on genomic differences and pursued differences in methylation patterns following CBT, but the findings were very limited in scope, especially when comparing responders and non-responders to CBT. In the currently proposed study, the investigators plan to go one step further and look for changes in exosomal microRNAs (miRs) from serum samples taken before and after CBT from Panic Disorder (PD) patients. Notably, miR changes show a much faster biological response than methylation patterns yet had never been used before in PD research. The primary benefit of this work will be in providing biological validation to psychological treatments. PD is a heavy public health burden, associated with significant market potential for both therapeutic and diagnostic uses.

DETAILED DESCRIPTION:
Cognitive Behavior Therapy (CBT) is an evidence-based treatment, commonly used for treating anxiety disorders. Patients with anxiety disorders are characterized by having cognitive distortions regarding evaluations of threat, which results in safety behaviors to avoid them thereby causing impairment in the patient's quality of life. CBT focuses on changing those "false beliefs" and "maladaptive behaviors" by exposing the patients to their anxiety source in a gradual way, supervised by the therapist.

Anxiety disorders are relatively common, and many people have difficulty accessing treatment due to a variety of obstacles. Researchers have therefore explored the possibility of using different methods to administer CBT, resulting in the making of internet-delivered CBT (iCBT). iCBT programs can involve therapist guidance through emails or can be entirely unguided. These programs are typically comprised of 6-15 modules, which are text chapters corresponding to sessions in face-to-face therapy. These programs require little therapist involvement other than guidance and feedback on homework assignments. Current meta-analyses suggest that iCBT does not differ from regular CBT in its efficacy, conducted through a guided program.

In this study, the investigators plan to examine whether iCBT and regular CBT can cause biological changes as well as cognitive ones. Few previous studies have shown epigenetic changes in different directions for CBT responders and non-responders. Those studies used methylation patterns as biomarkers, showing that Panic Disorder (PD) patients had lower methylation in specific genes than the control group at the baseline point. After going through CBT the responders showed higher methylation and the non-responders showed even lower methylation than at the baseline point. In addition, a more recent study showed that in comparison to healthy controls, PD patients showed changes in immune system activities. Microglial acid sensing G-protein coupled receptor and T cell death-associated gene-8 (TDAG8), which was found was found higher in PD patients.

The investigators wish to take these findings one step forward by using micro-RNAs (miRs) content of circulation exosomes as our biomarker. Exosomes are a type of extracellular vesicles of endocytic origin, used in signaling and cell to cell communication, by transferring proteins, lipids, and variety of RNAs between cells. miRs are short single-stranded RNA molecules that bind to complementary sequences of target mRNAs, causing inhibition of their translation and/or inducing target degradation and affecting brain functioning and mental processes.

The investigators will base their work on the hypothesis that the brain's state is reflected, to a certain extent in the miR contents of circulating exosomes. Therefore, the aim of the study will be to test the difference between patients and controls as well as between responders and non-responders by profiling miRs content of circulation exosomes from their plasma samples and seeking association with their clinical data. Whole blood samples will also be collected, in order to serve as secondary outcome measurement, checking for changes in expression of other small non-coding circulating RNAs as well.

The investigators will use a cohort of 40 panic disorder patients, comparing them with matching 40 mentally healthy controls. This approach has never been used before in the field of anxiety biomarkers, although miR changes show a much faster biological response than methylation patterns. Therefore, the investigators believe it will provide many new insights on the biological changes following PD and its treatment using CBT/iCBT, especially regarding the biological difference between respondents and non-respondents.

The investigators anticipate big benefits for psychologists and psychiatrists who could in the future use simple blood samples to determine which kind of therapy will be most suitable for their patients, or rather to check if the therapy has given the desirable outcomes. Biotech firms may be interested in developing this method as a commercial diagnostic tool that could easily be used by health maintenance organizations just as a simple blood test. PD is a big public health burden, leading the market potential both for therapeutics as well as diagnostics to be large in dollar terms.

This study received two ethics approvals that act together. The mentioned ethics approval given by the Hebrew university ethics committee was given for the psychological part of the experiment and include the CBT, using a psychologist or computer program. A second approval, Helsinki approval by the Hadassah hospital committee, covers the biological part of the experiment - including the blood drawing and further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Principal DSM-5 primary diagnosis of panic disorder and/or agoraphobia.
* Aged 18 years or older.
* PD duration of at least 3 months.
* If participant is on on medications for PD, the dosage has to remain constant for 3 months prior to the start of treatment and cannot be increased during treatment.
* The participant must have access to the internet and be willing to use it.

Exclusion Criteria:

* Substance abuse or dependence within the last 6 months.
* Active suicide potential within the last 6 months.
* Any current or history of psychosis or bipolar I disorder.
* Currently in weekly or biweekly psychotherapy.
* History of a complete course of panic focused CBT

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-03-24 (Actual); Primary Completion 2021-12-24 (Estimated); Study Completion 2021-12-24 (Estimated)

PRIMARY OUTCOMES:
Differntial expression of plasma exosomal microRNAs | Pre and post treatment, up to 6 months apart.
  Exosomes are a type of extracellular vesicles of endocytic origin, used in signalling and cell to cell communication, by transferring proteins, lipids, and variety of RNAs between cells. miRs are short single-stranded RNA molecules that bind to complementary sequences of target mRNAs, causing inhibition of their translation and/or inducing target degradation and affecting brain functioning and mental processes. Will be measured twice: pre and post treatment (post or 6 months, whichever is later, to the maximum of 6 months).

SECONDARY OUTCOMES:
Change in Panic Disorder Severity Scale (PDSS) | Weekly during treatment and at pre and post treatment evaluations, up to 6 months apart.
  Independent evaluators will conduct pre and post treatment evaluations and self report will be administered weekly. The PDSS can be administered as an interview or self-report measure. It is comprised of 7 items that are scored from 0-4, with a total scale score ranging from 0-28. Higher scores mean more severe panic disorder symptoms. Will be administered weekly during treatment, plus at pre and post treatment evaluations.
Change in Anxiety Sensitivity Index-3 (ASI-3) | Weekly during treatment and at pre and post treatment evaluations, up to 6 months apart.
  The ASI-3 is an 18-item self-report measure that measures beliefs regarding panic related bodily sensations. It will be used as a total score, which ranges from 0-72. The ASI-3 will be administered weekly. Higher scores mean more severe anxiety sensitivity.
Change in Mobility Inventory | Weekly during treatment and at pre and post treatment evaluations, up to 6 months apart.
  The Mobility Inventory is a self report measure of agoraphobic avoidance in which patients are asked to rate how much they avoid 26 situations on a 1-5 scale twice, once when alone and a second time when accompanied. The average score of all times will be used, which will range from 1-5. The MI will be administered weekly.
Differntial expression of whole Blood short non-coding RNAs | Pre and post treatment, up to 6 months apart.
  We will also collect whole blood samples that will serve as a secondary outcome measurement, checking for changes in expression of small non-coding circulating RNAs as well. This measurement will act as a more clinically accessible balance for the exosomes approach. Will be measured twice: pre and post treatment (post or 3 months, whichever is later, to the maximum of 6 months).
Change in the Five-Dimensional Curiosity Scale (DCS-5) | Pre and post treatment, up to 6 months apart.
  The DCS-5 is a self-report measure that measures 5 dimensions of curiosity via 25 items which are rated on a 1-7 scale. The total score of all 25 (ranging from 25-175) items and 5 subscales (each ranging from 5-35) will be used for this study. Will be measured twice: pre and post treatment (post or 6 months, whichever is later, to the maximum of 6 months).
Changes in Experiences in Close Relationship Scale-Short (ECR-s) | Pre and post treatment, up to 6 months apart.
  The ECR-s is a brief self report instrument that measures both Anxious and avoidance adult attachment styles. The two scales each contain 6 items rated on a 1-7 scale that are summed for each subscale, ranging from 6-42. Will be measured twice: pre and post treatment (post or 6 months, whichever is later, to the maximum of 6 months).
Changes in Sexual Functioning Questionnaire | Pre and post treatment, up to 6 months apart.
  this is a self-report measure of sexual functioning that is comprised of 14 items that are rated on a 1-5 scale and scored by a sum score that ranges between 14-70. Higher scores mean better sexual functioning. Will be measured twice: pre and post treatment (post or 6 months, whichever is later, to the maximum of 6 months).

CONTACTS AND LOCATIONS:
Overall Officials: Hermona Soreq, Professor, Principal Investigator — Hebrew University of Jerusalem; Ronen Segman, Professor, Principal Investigator — Hadassah Hebrew University Hospital; Salomon Israel, Professor, Principal Investigator — Hebrew University of Jerusalem
Locations (1):
- Hebrew University of Jerusalem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be placed on a public website after the manuscript is submitted for publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available once the manuscript is submitted for publishing.

REFERENCES:
- [Background] Alexander M, Hu R, Runtsch MC, Kagele DA, Mosbruger TL, Tolmachova T, Seabra MC, Round JL, Ward DM, O'Connell RM. Exosome-delivered microRNAs modulate the inflammatory response to endotoxin. Nat Commun. 2015 Jun 18;6:7321. doi: 10.1038/ncomms8321. PMID 26084661
- [Background] Andersson G, Cuijpers P, Carlbring P, Riper H, Hedman E. Guided Internet-based vs. face-to-face cognitive behavior therapy for psychiatric and somatic disorders: a systematic review and meta-analysis. World Psychiatry. 2014 Oct;13(3):288-95. doi: 10.1002/wps.20151. PMID 25273302
- [Background] Bekenstein U, Mishra N, Milikovsky DZ, Hanin G, Zelig D, Sheintuch L, Berson A, Greenberg DS, Friedman A, Soreq H. Dynamic changes in murine forebrain miR-211 expression associate with cholinergic imbalances and epileptiform activity. Proc Natl Acad Sci U S A. 2017 Jun 20;114(25):E4996-E5005. doi: 10.1073/pnas.1701201114. Epub 2017 Jun 5. PMID 28584127
- [Background] Barlow DH. Cognitive-behavioral therapy for panic disorder: current status. J Clin Psychiatry. 1997;58 Suppl 2:32-6; discussion 36-7. PMID 9078992
- [Background] Fruhbeis C, Helmig S, Tug S, Simon P, Kramer-Albers EM. Physical exercise induces rapid release of small extracellular vesicles into the circulation. J Extracell Vesicles. 2015 Jul 2;4:28239. doi: 10.3402/jev.v4.28239. eCollection 2015. PMID 26142461
- [Background] Huppert, J. D., & Baker-Morissette, S. L. (2003). Beyond the manual: The insider's guide to panic control treatment. Cognitive and Behavioral Practice, 10(1), 2-13.
- [Background] Meunier J, Lemoine F, Soumillon M, Liechti A, Weier M, Guschanski K, Hu H, Khaitovich P, Kaessmann H. Birth and expression evolution of mammalian microRNA genes. Genome Res. 2013 Jan;23(1):34-45. doi: 10.1101/gr.140269.112. Epub 2012 Oct 3. PMID 23034410
- [Background] Olthuis JV, Watt MC, Bailey K, Hayden JA, Stewart SH. Therapist-supported Internet cognitive behavioural therapy for anxiety disorders in adults. Cochrane Database Syst Rev. 2016 Mar 12;3(3):CD011565. doi: 10.1002/14651858.CD011565.pub2. PMID 26968204
- [Background] Roberts S, Lester KJ, Hudson JL, Rapee RM, Creswell C, Cooper PJ, Thirlwall KJ, Coleman JR, Breen G, Wong CC, Eley TC. Serotonin transporter [corrected] methylation and response to cognitive behaviour therapy in children with anxiety disorders. Transl Psychiatry. 2014 Sep 16;4(9):e444. doi: 10.1038/tp.2014.83. PMID 25226553
- [Background] Ziegler C, Richter J, Mahr M, Gajewska A, Schiele MA, Gehrmann A, Schmidt B, Lesch KP, Lang T, Helbig-Lang S, Pauli P, Kircher T, Reif A, Rief W, Vossbeck-Elsebusch AN, Arolt V, Wittchen HU, Hamm AO, Deckert J, Domschke K. MAOA gene hypomethylation in panic disorder-reversibility of an epigenetic risk pattern by psychotherapy. Transl Psychiatry. 2016 Apr 5;6(4):e773. doi: 10.1038/tp.2016.41. PMID 27045843
- [Background] Strawn JR, Mills JA, Sauley BA, Welge JA. The Impact of Antidepressant Dose and Class on Treatment Response in Pediatric Anxiety Disorders: A Meta-Analysis. J Am Acad Child Adolesc Psychiatry. 2018 Apr;57(4):235-244.e2. doi: 10.1016/j.jaac.2018.01.015. Epub 2018 Feb 8. PMID 29588049